CLINICAL TRIAL: NCT05953857
Title: " Knowing & Treating Kosaki/Penttinen Syndromes " International Collaborative Consortium. A Real-life Observational Study on the Natural History of KOGS and PS and on the Efficacy and Safety Profile of TKIs in These Patients.
Brief Title: Knowing and Treating Kosaki/Penttinen Syndromes
Acronym: IKKoPeS
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: OLIVIER-FAIVRE 2023
Record Dates: First submitted 2023-06-19; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Kosaki Overgrowth Syndrome; Penttinen Syndrome
MeSH Terms: conditions — Penttinen-Aula syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Untreated: Not treated with TKI
- Treated: Treated with TKI

SUMMARY:
Kosaki overgrowth syndrome (KOGS) and Penttinen syndrome (PS) are extremely rare multisystem disorders caused by heterozygous activating variants of the PDGFRB gene. KOGS results in characteristic craniofacial, orthopedic, skin and neurological disorders. PS is a progeroid disease responsible for a prematurely aged appearance. Patients suffer significant morbidity and mortality due to various complications. Tyrosine Kinase Inhibitors (TKIs) targeting PGDFRB appear to be a potential treatment option, as evidenced by a few case reports showing clinical improvement in some patients, with modest and self-resolving side effects. The natural history of these two syndromes remains poorly understood as only case-reports have been published.

Therefore, an international consortium was created in December 2019 by Pr FAIVRE (CHU Dijon Bourgogne & ERN ITHACA) to follow treated and untreated patients in a real-life, multicentre, observational study, in order to expand our knowledge of these ultra-rare diseases. In the longer term, we believe that TKIs could bring clinical benefit to KOGS/PS patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Kosaki or Penttinen syndrome
* Molecular diagnosis of an activating variant in PDGFRB gene
* Patient who has been informed and provide a written informed consent

Exclusion Criteria:

* Absence of clinical diagnosis of Kosaki or Penttinen syndrome
* Absence of molecular diagnosis of an activating variant in the PDGFRB gene.
* Patient who has not been informed and/or did not provide a written informed consent.

Ages: 0 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients with KOGS or PS due to PDGFRB activating variants
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2048-10 (Estimated)

PRIMARY OUTCOMES:
Symptom's burden | At various time points according to the type of symptom: from weekly to every 5 years
  Symptoms: type, severity, date of appearance, evolution

SECONDARY OUTCOMES:
Efficacy of TKI | Through the study completion, an average of 10 years.
  Proportion of patients with improvement in quality of life under TKI treatment, expressed as percentages
Safety of TKI | Through the study completion, an average of 10 years.
  Proportion of patients with side effects under TKI treatment, expressed as percentages
Percentage of patients whose follow-up complies with recommendations | Through the study completion, an average of 10 years.
Percentage of patients whose TKI has been chosen according to cellular studies | Through the study completion, an average of 10 years.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France